CLINICAL TRIAL: NCT07192744
Title: Rotigaptide in Endothelial Dysfunction?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: University of Aarhus (Other); University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Roti II
Record Dates: First submitted 2010-04-07; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Ischaemic Heart Diseases
Keywords: Ischaemia reperfusion; Gap junctions; Endothelial function
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): Ischaemia reperfusion (IR) injury (upper arm cuff inflated to 200 mmHg for 20 min) is induced during the study. Using bilateral forearm venous occlusion plethysmography, blood flow will be measured during intra-brachial infusion of acetylcholine (ACh; 5-20 µg/min) before and after IR injury and during intra-brachial co-infusion of saline-placebo
  Interventions: Procedure: Forearm vascular study
- 2 (Active Comparator): Ischaemia reperfusion (IR) injury (upper arm cuff inflated to 200 mmHg for 20 min) is induced during the study. Using bilateral forearm venous occlusion plethysmography, blood flow will be measured during intra-brachial infusion of acetylcholine (ACh; 5-20 µg/min) before and after IR injury and during intra-brachial co-infusion of rotigaptide
  Interventions: Procedure: Forearm vascular study

INTERVENTIONS:
Procedure: Forearm vascular study — Forearm blood flow measured by venous occlusion plethysmography during interarterial infusion of vasodilators (Ach). Venous blood sampling via cannula in antecubital fossa.

SUMMARY:
Arterial occlusion can lead to tissue ischemia and, if prolonged, end organ infarction. Clinical and experimental data would suggest that restoration of blood flow might trigger additional injury beyond that induced by the ischemia alone, so called Ischemia Reperfusion (IR) injury. IR injury impairs endothelial function through a mechanism that may involve intercellular gap junctions. Rotigaptide (ZP-123) is an anti-arrhythmic drug promoting intercellular coupling by increasing gap junction conductance. We intend to test the hypothesis that rotigaptide protects the forearm arterial circulation from IR-induced endothelial dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* healthy males between 18-65 years of ages, non-smokers.

Exclusion Criteria:

* Any concurrent illness or chronic medical condition. Concurrent use of vasoactive medication. Smoking history.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-09-19 (Actual); Primary Completion 2009-12-31 (Actual); Study Completion 2009-12-31 (Actual)

PRIMARY OUTCOMES:
Change in forearm blood flow after ischaemia reperfusion with or without co-infusion of Rotigaptide | 20 fixed timepoints throughout the study up to 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: David E Newby, PhD, FRCP, Study Director — University of Edinburgh; Rajesh K Kharbanda, PhD, FRCP, Study Director — University of Oxford
Locations (1):
- University of Edinburgh, 49 Little France Crescent, Edinburgh, United Kingdom